CLINICAL TRIAL: NCT06598085
Title: Clinical Trial Protocol to Evaluate the Efficacy and Safety of Laparoscopic Surgical Systems for Gynaecological Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cornerstone Robotics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F-00359-003
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06

CONDITIONS: Cervical Cancer; Endometrial Cancer
Keywords: Cervical Cancer; Endometrial Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot-assisted surgery (Experimental): Robot-assisted laparoscopic wide total hysterectomy
  Interventions: Device: Robot-assisted surgery

INTERVENTIONS:
Device: Robot-assisted surgery — Surgery with the Cornerstone Surgical Robot.

SUMMARY:
Evaluation of the efficacy and safety of thoracic and abdominal endoscopic surgical systems manufactured by Shenzhen Cornerstone Robotics Technology Co., Ltd. for use ingynaecological surgical procedures.

DETAILED DESCRIPTION:
The trial was designed using a prospective, single-centre, single-group target value approach.

For subjects who intend to undergo gynaecological surgery assisted by the Thoracic and Abdominal Endoscopic Surgical System.

To use the Thoracic and Abdominal Endoscopic Surgical System developed by Shenzhen Cornerstone Robotics Technology Co., Ltd. to perform surgery , and to evaluate the efficacy and safety of the experimental medical device in the surgical treatment

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years;
* Body Mass Height Index (BMI) 18<BMI<30kg/㎡;
* Patients identified by the investigator as suitable for general, gynaecological and thoracic surgery;
* Written informed consent.

Exclusion Criteria:

* Need for emergency surgery (e.g. gastric cancer, colorectal cancer combined with perforation, bleeding, obstruction, etc.);
* With other malignancies or a previous history of other malignancies.
* Preoperative imaging suggests that the tumour has distant metastases.
* The patient has a history of relevant surgery or previous history of other malignancy and is judged by the investigator to be unsuitable for enrolment.
* Severe bleeding tendencies or coagulopathic disorders.
* With long-term use of anticoagulant and anti-platelet drugs (anti-platelet aggregation drugs discontinued less than 1 week prior to surgery), history of bleeding disorders or hematopoietic or coagulation disorders.
* Significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or medication (e.g. systemic corticosteroids).
* With severe allergies and suspected or established alcohol, drug or substance addiction.
* Other conditions which, in the opinion of the investigator, make participation in this trial inappropriate.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Surgical non-referral rate | During the surgery
  Surgical untransferred is defined as not converted from an experimental medical device assisted method to another surgical device control system assisted, laparoscopic surgery or open surgery.

SECONDARY OUTCOMES:
The surgeon's operating time | During the surgery
  Operative time（minutes）
Intraoperative blood loss | During the surgery
  Estimated blood loss（milliliters，ml）
Length of postoperative stay | up to 12 weeks
  Total number of days the patient was in hospital from the day of surgery to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: JiangTao Fan, MD, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- Cornerstone Robotics, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tse KY, Ngan HYS, Lim PC. Robot-assisted gynaecological cancer surgery-complications and prevention. Best Pract Res Clin Obstet Gynaecol. 2017 Nov;45:94-106. doi: 10.1016/j.bpobgyn.2017.04.005. Epub 2017 Apr 23. PMID 28528932
- [Background] Pugin F, Bucher P, Morel P. History of robotic surgery: from AESOP(R) and ZEUS(R) to da Vinci(R). J Visc Surg. 2011 Oct;148(5 Suppl):e3-8. doi: 10.1016/j.jviscsurg.2011.04.007. Epub 2011 Oct 4. No abstract available. PMID 21974854
- See also: Ever since the US Food and Drug Administration approval of the use of da Vinci surgical systems (Intuitive Surgical Inc., Sunnyvale, California) in gynaecology in 2005, robot-assisted surgery has been widely adopted in different countries. — https://pubmed.ncbi.nlm.nih.gov/28528932/
- See also: History of robotic surgery: from AESOP® and ZEUS® to da Vinci® — http://pubmed.ncbi.nlm.nih.gov/21974854/